CLINICAL TRIAL: NCT01988545
Title: GLP-1's Influence on Intestinal Blood Flow
Brief Title: GLP-1's Effect on Cardiac Parameters and Mesenteric Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, MD ph.d. Lasse Bremholm, MD, ass. professor, ph.d, Zealand University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 2013.GLP-1
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: GLP-1; blood flow; cardiac out put; stroke volume; beat to beat; effect of GLP-1 on cardiac parameters and blood flow
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLP-1 (Active Comparator): 1,5 nmol/kg,GLP-1 sc injection
  Interventions: Other: 1,5 nmol/kg GLP-1 9-36amide, sc injection; Other: Exendin-4 ;10 ug,sc injection
- GLP-1 9-36amide (Active Comparator): 1,5 nmol/kg GLP-1 9-36amide, sc injection
  Interventions: Other: 1,5 nmol/kg,GLP-1 sc injection; Other: Exendin-4 ;10 ug,sc injection
- Exendin-4 (Active Comparator): Exendin-4 ;10 ug,sc injection
  Interventions: Other: 1,5 nmol/kg,GLP-1 sc injection; Other: 1,5 nmol/kg GLP-1 9-36amide, sc injection
- isotonic saline (Placebo Comparator): 2 ml of isotonic saline, sc injection
  Interventions: Other: 1,5 nmol/kg,GLP-1 sc injection; Other: 1,5 nmol/kg GLP-1 9-36amide, sc injection; Other: saline

INTERVENTIONS:
Other: 1,5 nmol/kg,GLP-1 sc injection
  Other Names: native GLP-1
  Arms: Exendin-4; GLP-1 9-36amide; isotonic saline
Other: 1,5 nmol/kg GLP-1 9-36amide, sc injection
  Arms: Exendin-4; GLP-1; isotonic saline
Other: Exendin-4 ;10 ug,sc injection
  Arms: GLP-1; GLP-1 9-36amide
Other: saline
  Arms: isotonic saline

SUMMARY:
to investigate the effect of the human incretin hormone GLP-1 on mesenteric blood flow and cardiac parameters

DETAILED DESCRIPTION:
to investigate the effect of the human incretin hormone GLP-1 on mesenteric blood flow and cardiac parameters, in healthy subjects, 4 arms, task force monitor

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* medical conditions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
blood flow | with in 120 minutes
  blood flow change measured by ultra sound

OTHER OUTCOMES:
cardiac parameters | with in 120 minutes
  measure of cardiac change with task force monitor

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Bremholm, MD, ph.d., Principal Investigator — Køge Hospital
Locations (1):
- Køge Hospital, Køge, State..., Denmark